CLINICAL TRIAL: NCT00583843
Title: Evaluation of Change in the Lumpectomy Cavity During Radiation Therapy by Weekly Ultrasound and by Daily Ultrasound During the Radiation Boost Dose
Brief Title: Ultrasound Targeting for the Lumpectomy Cavity
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jacobson, Geraldine M, Adjunct Clinical Professor, University of Iowa
Other Study IDs: 200602784
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Breast Neoplasms
Keywords: Lumpectomy; Ultrasonography; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ultrasound: The group of women who are being followed by Ultrasound.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound weekly during initial fields of radiation, and daily during the boost phase.

SUMMARY:
Accurate targeting of treatment sites should increase local control by radiation therapy for breast-cancer lumpectomy patients. Currently, ultrasound localization is used for prostate cancer patients to locate the prostate before daily radiation treatments. There is now documented evidence that the lumpectomy site does change during the external radiation therapy. Thus, treatment efficacy should be increased by localizing the target, monitoring volume changes, and adjusting the radiation target prior to the boost radiation dose.

DETAILED DESCRIPTION:
Study participants will have weekly ultrasounds performed of the lumpectomy cavity to determine shift and volume changed from the initial treatment-planning CT to the time of the radiation boost (approximately 4 weeks). These ultrasounds are done prior to their weekly doctor's appointment with Radiation Oncology.

When it is time to perform the radiation boost (when the radiation is more targeted to the lumpectomy cavity), the ultrasound will be done daily with the participant in treatment position. The SonArray system used for the ultrasound-driven targeting for prostate cancer will be utilized. If the lumpectomy cavity is observed, the ultrasound suggested shifts will be noted and compared to the shifts needed for standard clinical set up.

Once the subject has completed radiation therapy, the study participation is complete.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Patients must have histologically or cytologically confirmed breast carcinoma with voluntarily elected breast conservation techniques (i.e., lumpectomy)
* Age >18 years. Breast cancer, while not restricted only to adult women, is rare in the younger population.
* Radiation indicated as a post-surgical adjuvant treatment for breast conservation.
* Life expectancy of greater than 6 months.
* Karnofsky of greater or equal to 60
* The effects of radiation therapy on the developing human fetus at the recommended therapeutic dose can be abortifacient. For this reason, and because radiation therapy is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* The inability to visualize or reliably contour the lumpectomy cavity from the Radiation Oncology treatment planning CT scan.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the principal investigator.
* Pregnant women are excluded from this study because radiation therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with standard chemotherapeutic regimens (if applicable), breastfeeding should be discontinued if the mother is treated any adjuvant chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men who have had lumpectomy for the definitive treatment of breast cancer and have a defined cavity from this procedure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine the volume change in lumpectomy cavity during the course of external beam radiation prior to delivery of the radiation boost. | 7 weeks

SECONDARY OUTCOMES:
Determine by daily ultrasound if targeting of the CT-based boost field is inaccurate due to daily variation of subject position. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Jacobson, MD MPH, Principal Investigator — The Department of Radiation Oncology
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Jacobson G, Betts V, Smith B. Change in volume of lumpectomy cavity during external-beam irradiation of the intact breast. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1161-4. doi: 10.1016/j.ijrobp.2006.02.009. Epub 2006 May 6. PMID 16682143
- [Background] Warszawski A, Baumann R, Karstens JH. Sonographic guidance for electron boost planning after breast-conserving surgery. J Clin Ultrasound. 2004 Sep;32(7):333-7. doi: 10.1002/jcu.20050. PMID 15293299
- [Background] Gilligan D, Hendry JA, Yarnold JR. The use of ultrasound to measure breast thickness to select electron energies for breast boost radiotherapy. Radiother Oncol. 1994 Sep;32(3):265-7. doi: 10.1016/0167-8140(94)90026-4. PMID 7816945
- [Background] Leonard C, Harlow CL, Coffin C, Drose J, Norton L, Kinzie J. Use of ultrasound to guide radiation boost planning following lumpectomy for carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1993 Dec 1;27(5):1193-7. doi: 10.1016/0360-3016(93)90543-5. PMID 8262847